CLINICAL TRIAL: NCT06041789
Title: Effect of Acetylcholinesterase Inhibitors on Bone Metabolism and Fracture Risk Factors Among Older Adults With Mild to Moderate Alzheimer's Disease
Brief Title: Effect of Acetylcholinesterase Inhibitors on Bone Metabolism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00111080; R21AG078982 (NIH)
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Donepezil; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Donepezil (Experimental)
  Interventions: Drug: Donepezil
- Memantine (Active Comparator)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Donepezil — 10 mg tablet
  Arms: Donepezil
Drug: Memantine — 10 mg tablet
  Arms: Memantine

SUMMARY:
People with Alzheimer's disease are at an increased risk of bone fracture. Some studies have shown that those taking donepezil have a lower rate of bone fractures, but the reasons for this are unknown. The purpose of this study is to measure the effect of donepezil treatment on bone metabolism factors including bone mineral density, bone turnover markers, and bone quality.

Participants in this study will have a bone density test and have blood samples collected at the baseline study visit. Participants will then be randomly assigned to donepezil or matching memantine to be taken daily by mouth for 12 months. Blood samples will be collected at 6 and 12 months. A repeat bone density test will be performed at 12 months. Participants will also complete questionnaires at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cognitive impairment, including clinical assessment, radiographic or laboratory biomarker assessment
2. Willing to initiate treatment for cognitive impairment
3. A) For females: either age > 55 years, or Age < 55 years and at least 12 months since last menstrual period B) For males, age > 50 years
4. Geriatric Depression Scale score < 6
5. English-speaking

Exclusion Criteria:

1. Currently on acetylcholinesterase inhibitor or memantine
2. History of bradycardia, heart block, long QT, unexplained syncope, or other contraindication for donepezil; subject with ECG showing HR < 50, PR interval > 200 ms, QTc > 440 ms in men or > 460 ms in women, or evidence of atrioventricular block
3. Currently on osteoporosis medication (e.g., bisphosphonate, SERM, denosumab, teriparatide, abaloparatide, romozosumab, calcitonin)
4. Use of bisphosphonate within last 5 years
5. Use within last 6 months of estrogens or testosterone, androgen deprivation therapy or aromatase inhibitors, antiepileptic, heparin therapy, thiazolidinediones
6. History of disorders associated with secondary osteoporosis: collagen vascular diseases, malabsorption, inflammatory bowel disease, severe liver disease/cirrhosis, hyperthyroidism (endogenous or exogenous)
7. History of fracture of the humerus, wrist, or vertebra due to fall from standing height or less
8. History of hip fracture, hip replacement, or non-ambulatory
9. Long-term use (>6 months) of corticosteroids
10. History of Parkinson's, HIV, Huntington's disease
11. History of solid organ transplantation
12. History of bariatric surgery or intending to lose weight by bariatric surgery or weight loss medication (e.g. GLP-1 agonist) in the next 12-months
13. Severe kidney impairment (eGFR < 30 ml/min),
14. Active malignancy currently undergoing chemotherapeutic, surgical, or radiation therapy, except non-melanomatous skin cancer
15. 1-year mortality > 25%, measured by ePrognosis calculator
16. Planning to move out of the area in the next 12-months
17. Planning surgery in the next 12-months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in bone mineral density, as measured by dual x-ray absorptiometry (DXA) | baseline, 12 months

SECONDARY OUTCOMES:
Change in bone resorption marker C-terminal telopeptide (CTX) | baseline, 6 months, 12 months
  measured using commercially available ELISA test on serum
Change in bone formation marker amino-terminal propeptide of type I procollagen (P1NP) | baseline, 6 months, 12 months
  measured using commercially available ELISA test on serum
Change in Trabecular Bone score | baseline, 12 months
  measure of bone quality, using DXA spine images

CONTACTS AND LOCATIONS:
Overall Officials: Richard H Lee, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke Memory Disorders Clinic, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No